CLINICAL TRIAL: NCT00221312
Title: Alendronate to Prevent Perimenopausal Transition Bone Loss
Brief Title: Fosamax Bone Loss Study: Alendronate to Prevent Bone Loss
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Robert Jaffe, M.D., UCaliforniaSF
Other Study IDs: H675-20192; H675-20192-05; 39-62
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2005-05

CONDITIONS: Perimenopausal Bone Loss
Keywords: Perimenopausal bone loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fosamax

SUMMARY:
This is a study to determine if Fosamax (alendronate), a medication approved by the Food and Drug Administration (FDA) for the prevention and treatment of osteoporosis in postmenopausal women, is effective in decreasing the rate of bone loss which often begins to increase in the three to five years preceding the menopause (perimenopausal transition).

During the three to five years prior to the menopause, the rate of bone loss increases. One way that physicians treat this is with oral contraceptive medication. However, the incidence of complications from oral contraceptives after the age of 40 increases. Therefore, a non-hormonal means of preventing bone loss should be useful. Fosamax (alendronate) is in a class of compounds called bisphosphonates. This study is being done to determine whether Fosamax can be used to prevent the increased rate of bone loss during the perimenopausal transition.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 40-54 with symptomology of perimenopause including hot flashes, irregular periods and vaginal dryness.

Exclusion Criteria:

* Women should not be on hormone replacements, oral contraceptives, or bone mineral enhancing medications (bisphosphonates, selective estrogen receptor modulators [SERM's], parathyroid hormone [PTH], calcitriol, fluorides)
* They should not have any abnormalities of the esophagus which delay esophageal emptying
* They should not have hypocalcemia or severe kidney disease
* Their bone mineral density (T-score) should not be greater than 2 standard deviations.

Ages: 40 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Perimenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2002-05; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Jaffe, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States